CLINICAL TRIAL: NCT06237985
Title: Evaluation of the Effect of Conservative Root Canal Instrumentation on the Release of Inflammatory Mediators in Root Canal Treatments: a Randomized Clinical Trial
Brief Title: Effect of Conservative Root Canal Instrumentation on the Release of Inflammatory Mediators in Root Canal Treatments
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Sıla Nur Usta, Assistant Professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBU-GFOD-ENDO-SILANURUSTA-001
Record Dates: First submitted 2024-01-15; First posted 2024-02-02 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-01

CONDITIONS: Irreversible Pulpitis
Keywords: postoperative pain; endodontics; ELISA; conservative instrumentation
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Patients will be divided into 3 different file system randomly in order to measure the inflammatory mediators and postoperative pain.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients who will be treated and the assessor who will perform the analysis in lab will be blinded regarding which file is used for each patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ProTaper Gold file system (Experimental): Sx-S1-S2-F1-F2 files for mesial canals and F3 file for distal canal with 350 rpm speed and 2 Ncm torque will be used via an endodontic motor.
  Interventions: Procedure: ProTaper Gold file system
- OneShape file system (Experimental): 25/.06 file for mesial canals with 350 rpm and 4 Ncm torque will be used via an endodontic motor.
  Interventions: Procedure: OneShape file system
- TruNatomy file system (Experimental): 17/.02, 20/.04 ve 26/.04 files for mesial canals and 36/.03 file for distal canal with 500 rpm speed and 1.5 Ncm torque will be used via an endodontic motor.
  Interventions: Procedure: TruNatomy file system

INTERVENTIONS:
Procedure: ProTaper Gold file system — According to the manufacturers ' instructions, root canal treatments will be conducted with the ProTaper Gold rotary file system up to F2 for mesial canals.
  Arms: ProTaper Gold file system
Procedure: OneShape file system — According to the manufacturers ' instructions, root canal treatments will be conducted with the OneShape rotary file system up to 25/.06 for mesial canals.
  Arms: OneShape file system
Procedure: TruNatomy file system — According to the manufacturers ' instructions, root canal treatments will be conducted with the TruNatomy rotary file system up to 26/.04 for mesial canals.
  Arms: TruNatomy file system

SUMMARY:
The goal of this clinical trial is to evaluate the expression of inflammatory mediators in the crevicular fluid and periodontal ligament after one-visit root canal treatment of mandibular molars of patients with asymptomatic irreversible pulpitis using 3 different file systems.

The main question it aims to answer is: Does conservative root canal preparation cause decreased expression of inflammatory mediators compared to conventional root canal preparation?

In this context, patients will be divided into 3 groups based on the file systems as follows: ProTaper Gold, OneShape, and TruNatomy up to apical size #25. Both inflammatory mediator expression and postoperative VAS values will be compared.

DETAILED DESCRIPTION:
The below-mentioned steps will be performed in the scope of this study:

1. Ethical approval has been obtained.
2. The sample size calculation was performed (90% power, 0.597 effect size, 20 patients per group)
3. Patients aged 18-60 with asymptomatic irreversible pulpitis that has been confirmed by intraoral and extraoral examination and without any systemic disease will be included.
4. Only mandibular first and second molar teeth that do not have complex anatomy, periapical lesions, deep periodontal pockets (PAI<2), and any fractures or cracks will be included.
5. Patients with acute symptoms, a history of taking analgesics 48 hours or antibiotics within 1 month prior to the visit, being pregnant and lactating, and having several periodontal problems will be excluded.

5) Immature apexes and trauma cases will also be excluded. 6) Selected patients will be informed about the study, and written consent will be obtained from all patients.

7) Patients will be randomly distributed into groups using a software (www.randomizer.org). Moreover, patients will be blinded regarding the file system they use.

8) A single operator will perform all endodontic treatments in the same clinical conditions.

9) Before starting the treatment, the baseline Visual Analogue Scale (VAS) values will be recorded.

10) For baseline inflammatory mediator assessment, gingival crevicular fluid samples from mesial and distal surfaces from teeth with #20 paper points for 30 seconds and paper points will be placed into Eppendorf tubes and kept at -80 ° until the analysis is performed.

11) After the administration of the local anaesthesia, teeth will be isolated with a rubber dam, and access cavities will be prepared. Then, teeth will be allotted to one of the following file systems:

* Group 1 (ProTaper Gold file system): Sx-S1-S2-F1-F2 (for mesial canals), F3 (for distal canal)
* Group 2 (OneShape file system): 25/.06 (for mesial canals), additional file for distal canal if needed.
* Group 3 (TruNatomy file system): 17/.02, 20/.04 ve 26/.04 (for mesial canals), 36/.03 (for distal canal.)

  12) 2 mL 2.5% sodium hypochlorite (NaOCl) will be used between files and final irrigation will be performed using 5 mL NaOCL, 5 mL 17% ethylenediaminetetraacetic acid (EDTA), and 5 mL distilled water with 31-G side vented needle.

  13) After drying the canals, #15 paper point will be placed inside mesial canals for 1 minute, 2 mm beyond the apex. Afterwards, paper points will be placed into Eppendorf tubes and kept at -80 ° until the analysis is performed.

  14) Root canals will be obturated with resin-based sealer and gutta-percha. 15) Permanent restoration will be done using composite. 16) Patients will be recalled at 24 and 72 hours, and gingival crevicular fluid samples from mesial and distal surfaces will be obtained using an above-mentioned method.

  17) Measurement of postoperative pain after treatment with a VAS scale at 24, 48, and 72 hours will also be recorded.

  18) Measurement of pain mediators (Substance P, Prostaglandin E2, interleukin (IL) 6, and IL-10) will be performed with ELISA kits. All samples will be analyzed in duplicate.

  19) Based on the readings obtained from the spectrophotometer, results will be fitted to the standard curve and presented in the form of picograms per millilitre (pg/mL).

  20) Statistical analysis will be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-60
* Patients with asymptomatic irreversible pulpitis that has been confirmed by intraoral and extraoral examination
* Patients with pain pain between 0 and 3 on the VAS scale
* Patients without any systemic disease
* Mandibular first and second molar teeth without complex root canal anatomy, calcifications, periapical lesions, deep periodontal pockets (PAI<2), and any fractures or cracks

Exclusion Criteria:

* Patients with acute symptoms
* Patients who have a history of taking analgesics 48 h or antibiotics within 1 month prior to the visit
* Patients who are being pregnant and lactating
* Patients with several periodontal problems
* Patients with systemic disease
* Teeth with immature root apexes
* Trauma cases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Measurement of Substance P | Before root canal treatment (Day 0), at 24 hours, and at 72 hours
  Measurement of Substance P
Measurement of Prostaglandin E2 | Before root canal treatment (Day 0), at 24 hours, and at 72 hours
  Measurement of Prostaglandin E2
Release of inflammatory mediators | Before root canal treatment (Day 0), at 24 hours, and at 72 hours
  Measurement of Prostaglandin IL-6
Measurement of IL-10 | Before root canal treatment (Day 0), at 24 hours, and at 72 hours
  Measurement of IL-10

SECONDARY OUTCOMES:
Postoperative pain assessment using visual analog scale | Before root canal treatment (Day 0), at 24 hours, and at 72 hours
  Postoperative pain assessment using visual analog scale

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Karaoğlanoğlu, Professor, Study Director — Saglik Bilimleri Universitesi

IPD SHARING:
Plan to Share IPD: No
Within the scope of the necessity of protecting the individual information of the patients, it is considered that the recorded data will not be shared.

REFERENCES:
- [Result] Kasikci S, Turker SA, Guven B. Effect of different retreatment files using different kinematics on the release of inflammatory mediators in root canal retreatment of single-rooted teeth: a randomized clinical trial. Clin Oral Investig. 2023 Jun;27(6):3189-3196. doi: 10.1007/s00784-023-04930-6. Epub 2023 Mar 1. PMID 36856848
- [Result] Bicakci H, Capar ID, Genc S, Ihtiyar A, Sutcu R. Influence of Rotary Instrumentation with Continuous Irrigation on Pain and Neuropeptide Release Levels: A Randomized Clinical Trial. J Endod. 2016 Nov;42(11):1613-1619. doi: 10.1016/j.joen.2016.08.010. PMID 27788771
- [Result] Nunez N, Erdogan O, Casey SM, Hernandez R, Tan S, Gibbs JL. Elevated Cytokine Levels in Gingival Crevicular Fluid of Teeth with Apical Periodontitis. J Endod. 2023 Jun;49(6):657-663. doi: 10.1016/j.joen.2023.03.010. Epub 2023 Mar 24. PMID 36965768
- [Result] Shin SJ, Lee W, Lee JI, Baek SH, Kum KY, Shon WJ, Bae KS. Matrix metalloproteinase-8 and substance P levels in gingival crevicular fluid during endodontic treatment of painful, nonvital teeth. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2011 Oct;112(4):548-54. doi: 10.1016/j.tripleo.2011.04.026. Epub 2011 Aug 10. PMID 21831678
- [Result] Canakci BC, Er O, Genc Sen O, Sut N. The effect of two rotary and two reciprocating NiTi systems on postoperative pain after root canal retreatment on single-rooted incisor teeth: A randomized controlled trial. Int Endod J. 2021 Nov;54(11):2016-2024. doi: 10.1111/iej.13609. Epub 2021 Aug 29. PMID 34383324